CLINICAL TRIAL: NCT06848244
Title: Preventing Type 2 Diabetes in Black Emergent Adult Women At-Risk for Binge-Eating Disorder
Brief Title: Preventing Type 2 Diabetes in Black Emergent Adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 25-0125
Record Dates: First submitted 2025-02-14; First posted 2025-02-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus; Binge-Eating Disorder; Binge Eating; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Binge-Eating Disorder; Bulimia; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appetite Awareness Training (AAT) and Diabetes Prevention Program (DPP) (Experimental): Participants are randomized into the AAT and DPP groups and receive content from both programs for 12 months.
  Interventions: Behavioral: Appetite Awareness Training (AAT); Behavioral: Diabetes Prevention Program (DPP)
- Diabetes Prevention Program (DPP) only (Experimental): Participants are randomized into the DPP group and will be able to access the program's content.
  Interventions: Behavioral: Diabetes Prevention Program (DPP)

INTERVENTIONS:
Behavioral: Appetite Awareness Training (AAT) — Partcipants will receive the AAT delivered as 16 core sessions over six months as well as six maintenance sessions over the course of 12 months.
  Arms: Appetite Awareness Training (AAT) and Diabetes Prevention Program (DPP)
Behavioral: Diabetes Prevention Program (DPP) — Partcipants will receive the DPP delivered as 16 core sessions over six months as well as six maintenance sessions over the course of 12 months.

SUMMARY:
Black Americans are disproportionately affected by diabetes, with nearly double the rates of type 2 diabetes mellitus (T2DM), compared to non-Hispanic White adults. Though numerous factors affect these disparities, one modifiable risk factor may be that of binge eating (BE), which increases risk for binge-eating disorder (BED), which is associated with severe obesity, and often precedes a T2DM diagnosis, beginning in childhood or adolescence. Nearly 30% of Black women with obesity report binge eating episodes. Furthermore, given that binge and overeating may disparately increase the odds of obesity in Black adults (15-fold increase vs. 6-fold increase in White adults), reducing this behavior will be critical to prevent continued disparities in T2DM diagnosis. Given that Black women have the highest rates of obesity in the nation (57%), report disparate rates of weight gain between young adulthood and mid adulthood, and report disparate rates of emotional eating in adolescence, which is a risk factor for BE, one pathway to reducing disparities in T2DM risk in Black women may be to reduce binge eating and prevent weight gain in emerging adulthood (ages 18-25).

DETAILED DESCRIPTION:
Aim 1. Use formative research to gather recommendations to Tailor AAT+DPP to Black Emergent Adult (EA) Women (Year 1).

Aim 2. Utilize community-engaged and user-centered design methods to adapt a mobile intervention to prevent T2DM in Black women at risk for BED (Year 2).

Aim 3. Conduct a pilot randomized trial to examine the feasibility and acceptability, and preliminary efficacy of the adapted AAT+ DPP intervention (Years 3-4; Analysis Year 5).

ELIGIBILITY:
Inclusion Criteria:

* Black women
* between 18-25 years of age
* BMI ≥ 25 kg/m^2
* At least one binge eating episode weekly
* Prediabetic
* Have access to a smartphone

Exclusion Criteria:

* Have no internet access
* Currently type 2 diabetic
* Currently pregnant
* Are in substance use treatment
* Have received prior or planned bariatric surgery

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of Binge Eating Episodes from Baseline to Month 6 | Baseline, 6 months
  Participants will self-monitor and complete surveys on binge eating episodes.
Change from Baseline to Month 6 in weight regain | Baseline, 6 months
  Participant body weight will be measured by trained research staff using calibrated digital scales. Participants will be in light indoor clothing, with pockets emptied, and belts and shoes removed.

SECONDARY OUTCOMES:
Change in Inflammatory Biomarkers for T2DM from Baseline to Month 6 | Baseline, 6 months
  Participants will provide plasma samples to examine the risk for type 2 diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Goode, PhD,MPH,LCSW, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No